CLINICAL TRIAL: NCT00181818
Title: Safety and Efficacy of Sustained-Release (SR) Bupropion for Smokers Hospitalized Smokers With Acute Coronary Heart Disease
Brief Title: Bupropion for Hospitalized Smokers With Acute Cardiovascular Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1999-P-002639; NIH: R01 HL61779
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-09

CONDITIONS: Smoking; Myocardial Infarction; Unstable Angina; Cardiovascular Disease
Keywords: Smoking cessation; Bupropion SR; Hospital intervention; Myocardial infarction; Unstable angina
MeSH Terms: conditions — Smoking; Myocardial Infarction; Angina, Unstable; Cardiovascular Diseases; Smoking Cessation

INTERVENTIONS:
Drug: bupropion SR (sustained-release)

SUMMARY:
The purpose of the study is to test the efficacy and safety of bupropion SR for smokers hospitalized with acute cardiovascular disease.

DETAILED DESCRIPTION:
Each year, over 2 million Americans are hospitalized with a myocardial infarction (MI) or unstable angina pectoris, two acute and potentially fatal manifestations of coronary heart disease (CHD). Smoking cessation is highly cost-effective and universally recommended for the approximately 20% of these patients who smoke. Hospitalization for acute CHD is an excellent time to initiate smoking cessation because hospitalization requires temporary tobacco abstinence at the same time that illness increases smokers' motivation to quit. Unfortunately, at least 40% of smokers fail to quit even with optimal cognitive-behavioral counseling interventions that begin in the hospital and continue after discharge. More powerful intervention strategies are needed. Adding pharmacotherapy to behavioral counseling, which is standard practice in outpatients, has not been tested in this setting because of concern about the safety of nicotine replacement after MI. Sustained release (SR) bupropion (Zyban, Wellbutrin SR) is a non-nicotine antidepressant drug that has recently proved to be effective for smoking cessation. It appears to be safe in cardiac patients and may have the additional benefit of preventing post-MI depression, an independent predictor of mortality.

This study tested the efficacy and safety of bupropion SR for smoking cessation in adult smokers hospitalized with MI or unstable angina. To do so, we conducted a five-site randomized double-blind placebo-controlled trial to determine whether bupropion SR, initiated in the hospital and continued for 12 weeks, was effective and safe when added to comprehensive cognitive-behavioral smoking counseling. The primary outcome measure was biochemically-confirmed 7-day point prevalence tobacco abstinence at 1 year follow-up. Principal secondary outcome measure was biochemically-confirmed 7-day point-prevalence at end-of-treatment (12 weeks). Secondary aims were to test whether bupropion SR delays the time to smoking relapse, reduces CHD morbidity and depressive symptoms, and improves health-related quality of life over 1 year of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old,
* had smoked >1 cigarette in the past month,
* were admitted to the hospital with a diagnosis of acute cardiovascular disease (see below)
* had an expected hospital stay of >24 hours.

Eligible admission diagnoses included (1) acute ischemic coronary heart disease (MI or unstable angina), (2) coronary artery bypass graft surgery, or (3) other cardiovascular conditions (congestive heart failure, cardiac arrhythmia, valvular heart disease, or atherosclerotic disease of the aorta, carotid, renal or peripheral arteries) in subjects with documented coronary artery disease.

Exclusion Criteria:

* not willing to consider smoking cessation after discharge,
* a contraindication to bupropion (seizure disorder, monoamine oxidase inhibitor use, history of anorexia nervosa or bulimia, bupropion allergy)
* a condition that increased the risk of seizure (e.g., serious head trauma with loss of consciousness
* uncontrolled hypertension (BP >160/100) in hospital
* heavy alcohol use (>3 drinks/day) or binge drinking (>6 drinks for males or >5 drinks for females) at least monthly
* renal insufficiency (serum creatinine >2.0 mg/dl),
* severe hepatic disease
* severe depression or severe cognitive impairment or psychosis
* life expectancy of <12 months,
* illegal drug use in the past 6 months
* bupropion use in the past month
* non-English speaking
* no telephone
* residence outside a defined geographic area.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248
Dates: Start 1999-10; Study Completion 2003-12

PRIMARY OUTCOMES:
Cotinine-validated 7-day point prevalence tobacco abstinence at 1 year follow-up
Cotinine-validated 7-day point prevalence tobacco abstinence at 3 month follow-up (end of treatment)

SECONDARY OUTCOMES:
Combined fatal and nonfatal cardiovascular events at 3 month follow-up (end of treatment)
Combined fatal and nonfatal cardiovascular events at 1 year follow-up
Cardiovascular mortality at 1 year follow-up
Blood pressure elevation (SBP>160 or DBP>100) during treatment with study drug

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961
- [Derived] Thorndike AN, Regan S, McKool K, Pasternak RC, Swartz S, Torres-Finnerty N, Rigotti NA. Depressive symptoms and smoking cessation after hospitalization for cardiovascular disease. Arch Intern Med. 2008 Jan 28;168(2):186-91. doi: 10.1001/archinternmed.2007.60. PMID 18227366
- [Derived] Rigotti NA, Thorndike AN, Regan S, McKool K, Pasternak RC, Chang Y, Swartz S, Torres-Finnerty N, Emmons KM, Singer DE. Bupropion for smokers hospitalized with acute cardiovascular disease. Am J Med. 2006 Dec;119(12):1080-7. doi: 10.1016/j.amjmed.2006.04.024. PMID 17145253